Official Title: A Randomized Controlled Trial of Vitamin D Supplementation in Multiple Sclerosis

NCT01490502

March 14, 2022

# **Statistical Analysis Plan**

- I. Title: The vitamin D to ameliorate multiple sclerosis (VIDAMS) trial: Statistical Analysis Plan
- II. Trial Manuscript Leadership Team: Ellen M. Mowry, MD, MCR (PI) and Sandra D. Cassard, ScD (Co-I, manuscript lead)
- III. Statistician: Kathryn C. Fitzgerald, ScD
- IV. Intervention
  - a. Low dose vitamin D₃ supplementation (LDVD) of 600 IU/day + glatiramer acetate
  - b. High dose vitamin D₃ supplementation (HDVD) of 5000 IU/day + glatiramer acetate
- V. Outcomes:
  - a. Primary outcome (clinical outcome)
    - i. Proportion of participants who experienced a confirmed relapse
  - b. Secondary outcomes (separated out to clinical and radiographic)
    - i. Clinical outcomes:
      - 1. Confirmed or probable relapse
      - 2. Annualized relapse rate
      - 3. Number of relapses requiring treatment
      - 4. Sustained disability progression
        - a. Defined as change in EDSS scores at 1 year that was sustained at year 2. Progression is defined as an increase in EDSS score of 1.0.
          - i. Use screening rather than baseline EDSS to compute change if relapse between screening and baseline.
      - 5. Change in multiple sclerosis (MS) functional composite (MSFC)
        - a. Change in components of MSFC. These include walking speed, 9-hole peg test, and PASAT-3.
        - b. MSFC will be considered as a Z score; MSFC component tests will be assessed as raw and Z scores.
        - c. Sustained 20% worsening from baseline MSFC that is confirmed at a subsequent visit.
      - 6. Change in low contrast letter acuity (LCLA)
        - a. Raw change in number of correct letters
        - b. Sustained 20% worsening from baseline LCLA that is confirmed at a subsequent visit.
        - c. Sustained change of ≥7 letter (clinically meaningful change)
      - 7. Change in health-related quality of life using the functional assessment in MS (FAMS) scores
        - a. These include the total FAMS score and components for symptoms, mobility, fatigue, emotional well-being, social well-being
        - b. 0.5 SD improvement in FAMS total and component scores
      - 8. Development of hypercalcemia and other adverse events
        - a. Hypercalcemia is defined as serum calcium level 0.5 mg/dL above the upper limit of normal; severe hypercalcemia is defined as ≥1 mg/dL above the upper limit of normal.
        - b. Self-reported development of kidney stones at any time during follow-up.
    - ii. MRI outcomes:
      - 1. T2 lesion volume
      - 2. Number of new/enlarged T2 lesions
      - 3. Number of Gadolinium enhancing (Gd+) lesions
      - 4. Composite sum of number of new lesions (sum of Gd+ and new/enlarged T2 lesions)
      - 5. Proportion developing a new lesion over follow-up.
      - 6. Normalized brain parenchymal fraction (nBPV)
      - 7. Normalized gray matter volume (nGMV)
      - 8. Normalized white matter volume (nWMV)

### VI. Descriptive Analyses

a. Characterize baseline cohort overall and by randomization arm for demographic, clinical, and patient characteristics in a table with 3 columns (overall, LDVD, HDVD) using descriptive statistics based on the variable in question (e.g., means and standard deviations, median and interquartile range, and percentages).

- i. These characteristics will be included: age, sex, race, ethnicity, disease subtype (relapsing remitting MS vs. clinically isolated syndrome), body mass index (BMI), previous treatment with a MS disease modifying therapy (DMT), EDSS scores, T2 lesion volume, skin tone, and sun exposure, nBPV, nGMV, and nWMV
- b. Characterize 25-hydroxyvitamin D (25[OH]D) levels overall and by randomization arm at baseline and over time (screening, baseline, and months 3, 6, 12, 18, and 24)
  - i. Characterize missing data in 25(OH)D levels by randomization arm and by time
  - ii. Calculate descriptive statistics for 25(OH)D levels by randomization arms and by time.
  - iii. Plot means (SD) of 25(OH)D levels by randomization arm over time
  - iv. Create spaghetti plots with overlaid loess curves for 25(OH)D levels by randomization arm over time.
  - v. Plot 25(OH)D levels by season (or month) of blood draw and by randomization arm and time to confirm no differences.
  - vi. Plot 25(OH)D levels by region of blood draw and by randomization arm and time to confirm no differences.

# VII. Consort Diagram

a. A consort diagram will be created with the following levels: assessed for eligibility, randomized, treatment allocation, follow-up and analytic cohort.

## VIII. Regression models: Intention to treat analyses

- a. We will incorporate variables with differences between the treatment arms that exceed 10% as identified using results of the descriptive analyses (e.g., sex, race, or ethnicity).
- b. Eligible participants for the primary analysis are those with baseline data and at least one follow-up visit.
- c. Missing values for key baseline covariates of interest is expected to be small; however, primary analyses will include a missing indicator level for the categorical variable if it is included in analytic models. The sensitivity of results will be assessed using pattern mixture models<sup>1</sup> and shared random effects models.<sup>2</sup>
- d. For mixed effects models, time will be considered as a linear variable in primary analyses. Secondary analyses will account for time as a categorical variable.
- e. Primary outcome: proportion of individuals with a relapse.
  - i. Proportion with a confirmed relapse will be assessed using a Cox proportional hazards model to account for follow-up time and accounting for identified potentially unbalanced covariates
  - ii. Plot unadjusted results using Kaplan Meier curves and test for significance using log-rank test (or other appropriate test if assumptions are not met for log-rank).

# f. Secondary outcome:

- i. Clinical outcomes
  - 1. Proportion with a confirmed or probable relapse
    - a. Proportion with a confirmed or probable relapse will be assessed using a Cox proportional hazards model to account for follow-up time
  - 2. Annualized relapse rate (two sets: confirmed, confirmed or probable)
    - a. Using an Andersen-Gill model for time to recurrent events correcting for dependence between multiple events assess risk of MS relapse
    - b. Plot unadjusted results using Kaplan Meier curves and test for significance using log-rank test (or other appropriate test if assumptions are not met for log-rank).
  - 3. Number of relapses requiring treatment
    - a. Using a negative binomial model incorporating follow-up time using as an offset term. Results will be presented as rate ratio estimates comparing HDVD vs. LDVD.
  - 4. Sustained disability progression
    - a. Using a Cox proportional hazards model
    - b. Plot unadjusted results using Kaplan Meier curves and test for significance using log-rank test (or other appropriate test if assumptions are not met for log-rank).
  - 5. Change in multiple sclerosis (MS) functional composite (MSFC)
    - a. Rate of change in MSFC Z scores (and component Z scores) using a linear mixed effects model with unstructured covariance structure, random intercepts. If model fit is improved with the addition of random slopes, they will be added.

- b. Rate of change in raw components using a linear mixed effects model with unstructured covariance structure, random intercepts. If model fit is improved with the addition of random slopes, they will be added. A log transformation will be applied if data are skewed based on visual inspection.
- c. For 20% change models, we will fit statistical models if ≥10 events occurred. Time to 20% worsening in MSFC (and components) using a Cox proportional hazards model.
- d. Plot unadjusted results using Kaplan Meier curves for time to event outcomes and test for significance using log-rank test (or other appropriate test if assumptions are not met for logrank).

# 6. Change in LCLA

- a. Rate of change in LCLA using a linear mixed effects model with unstructured covariance structure, random intercepts. If model fit is improved with the addition of random slopes, they will be added.
- b. For 20% change and 7-letter change models, we will fit statistical models if ≥10 events occurred. Time to 20% worsening or 7-letter loss in LCLA will be assessed using a Cox proportional hazards model.
- c. Plot unadjusted results using Kaplan Meier curves for time to event outcomes and test for significance using log-rank test (or other appropriate test if assumptions are not met for log-rank).
- 7. Change in health-related quality of life using the functional assessment in MS (FAMS) scores
  - a. Rate of change in quality of life using a linear mixed effects model with unstructured covariance structure, random intercepts. If model fit is improved with the addition of random slopes, they will be added.
  - b. For ≥ 0.5 SD improvement, we will fit statistical models if ≥10 events occurred. Time to ≥ 0.5 SD improvement in FAMS total score and subscale scores will be assessed via Cox proportional hazards model.
  - c. Plot unadjusted results using Kaplan Meier curves and test for significance using log-rank test (or other appropriate test if assumptions are not met for log-rank).
- 8. Development of hypercalcemia adverse events
  - a. Proportion of patients developing hypercalcemia or kidney stones will be compared descriptively
  - b. A logistic regression model will be considered if the number of events for either adverse event exceeds 10.

### ii. MRI outcomes:

- 1. T2 lesion volume
  - a. Rate of change in T2 lesion volume using a linear mixed effects model with unstructured covariance structure, random intercepts. If model fit is improved with the addition of random slopes, they will be added.
- 2. Number of new/enlarged T2 lesions
  - a. Using a negative binomial model incorporating follow-up time using as an offset term.
- 3. Number of Gadolinium enhancing (Gd+) lesions
  - a. Using a negative binomial model incorporating follow-up time using as an offset term.
- 4. Composite number of new lesions (sum of Gd+ and new/enlarged T2 lesions)
  - a. Using a negative binomial model incorporating follow-up time using as an offset term.
- 5. Proportion developing a new lesion
  - a. Proportion developing a new lesion will be assessed using a Cox proportional hazards model to account for follow-up time and accounting for identified potentially unbalanced covariates
  - b. Plot unadjusted results using Kaplan Meier curves and test for significance using log-rank test (or other appropriate test if assumptions are not met for log-rank).

### 6. nBPV

a. Rate of change in nBPV using a linear mixed effects model with unstructured covariance structure, random intercepts. If model fit is improved with the addition of random slopes, they will be added.

### 7. nGMV

a. Rate of change in nGMV using a linear mixed effects model with unstructured covariance structure, random intercepts. If model fit is improved with the addition of random slopes, they will be added.

### 8. nWMV

 Rate of change in nWMV using a linear mixed effects model with unstructured covariance structure, random intercepts. If model fit is improved with the addition of random slopes, they will be added.

## IX. Regression models: Planned per protocol analyses

- a. For planned per protocol analyses, we will consider the following analyses for the primary outcome proportion with a confirmed relapse and secondary outcomes including proportion with a confirmed or probable relapse, annualized relapse rate, proportion developing a new lesion, change in overall MSFC Z score.
- b. Overview of planned per-protocol analyses
  - i. Accounting for change in disease modifying therapy using the following models:
    - 1. DMTs will be included as a time-varying covariate in Cox models.
    - 2. Individuals will be censored upon switching DMTs
    - 3. Inverse probability weighted models account for therapy changes; weights analysis will also incorporate premature censoring (see iv).
  - ii. Assessing differences by adherence to study medication or drug
    - 1. Patient adherence to treatment will be included as a time-varying covariate; the variable will be derived using all available information (missed doses, pill counts).
      - a. Likely to categorize to deal with heterogeneity in collection of data
      - b. Missing carried forward
    - 2. Patient adherence to MS DMTs will be included as a time-varying covariate using self-reported patient medication adherence.
  - iii. Mediation by change in 25(OH)D levels
    - 1. The effect of change in 25(OH)D on primary outcomes will be assessed using instrumental variables and 2-stage residual inclusion with study-group assignment as the instrument and change in 25(OH)D level from baseline as the exposure of interest.<sup>3</sup>
  - iv. Assessing predictors of drop-out/early censoring
    - 1. Baseline covariates will be used to assess whether certain characteristics were associated with follow-up time.
    - 2. Sensitivity analyses will fit inverse probability weighted models accounting for premature censoring or therapy changes (as in i).
  - v. Determination of treatment response scores to quantify predictors of participants who will respond "responders"
    - 1. Treatment response scores will be derived using baseline participant characteristics to assess and quantify potential heterogeneous treatment effects<sup>4–6</sup>
  - vi. Assessing whether inclusion of individuals with high inflammatory activity impact the results.
    - 1. A person with high inflammatory activity is defined as individuals with ≥4 relapses over the study period.
    - 2. Check the distribution for Gd+ enhancing lesions at baseline and over follow-up. If clear outliers (>+4SD) then analyses excluding these individuals.
  - vii. Assessing effect modification by skin tone using Fitzpatrick scale and sun exposure
    - 1. Stratified analyses will assess effect modification by skin tone and sun exposure.

### References

- 1. Little RJA. Pattern-Mixture Models for Multivariate Incomplete Data. Journal of the American Statistical Association 1993;88(421):125–134.
- 2. Follmann D, Wu M. An Approximate Generalized Linear Model with Random Effects for Informative Missing Data. Biometrics 1995;51(1):151–168.

- 3. Terza JV, Basu A, Rathouz PJ. Two-stage residual inclusion estimation: Addressing endogeneity in health econometric modeling. Journal of Health Economics 2008;27(3):531–543.
- 4. Bovis F, Carmisciano L, Signori A, et al. Defining responders to therapies by a statistical modeling approach applied to randomized clinical trial data. BMC Med 2019;17(1):113.
- 5. Zhao L, Tian L, Cai T, et al. EFFECTIVELY SELECTING A TARGET POPULATION FOR A FUTURE COMPARATIVE STUDY. J Am Stat Assoc 2013;108(502):527–539.
- 6. Pellegrini F, Copetti M, Bovis F, et al. A proof-of-concept application of a novel scoring approach for personalized medicine in multiple sclerosis. Mult Scler 2020;26(9):1064–1073.